CLINICAL TRIAL: NCT00898222
Title: Effect of Daily Low Dose Aspirin on Exhaled Inflammatory Mediators in Normal Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Elliot Israel, MD, Elliot Israel, MD, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ARC ASA Normal
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Results first posted 2014-11-04 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: healthy volunteers; aspirin; Normal healthy subjects
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- aspirin (Experimental): Low dose daily aspirin in healthy volunteers for two weeks
  Interventions: Drug: aspirin

INTERVENTIONS:
Drug: aspirin — 81 mg orally daily for two weeks

SUMMARY:
Hypothesis: Low dose aspirin does not change exhaled inflammatory breath mediators in normal subjects.

DETAILED DESCRIPTION:
Aim:

1. To study the effect of low dose aspirin on exhaled breath inflammatory mediators
2. To compare the change to that seen in diseased states such as asthma and Lymphangioleiomyomatosis (LAM)

We will interview healthy volunteers to confirm that they do not have any major underlying medical conditions such as heart disease, diabetes, stroke and bleeding disorders. We will collect breath condensate before and after two weeks of low dose over the counter enteric coated aspirin 81 mg/day therapy. Side effects are extremely rare at this dose, but include bleeding, heart burn and allergic reaction.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults

Exclusion Criteria:

* any underlying major medical conditions such as heart disease, hypertension, stroke, diabetes, bleeding disorders

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shamsah Kazani, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Asthma Research Center, Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Aspirin: Low dose daily aspirin in healthy volunteers for two weeks
  aspirin : 81 mg orally daily for two weeks
Period: Overall Study
Arm/Group | Aspirin
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Aspirin
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (2.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Exhaled Inflammatory Mediator Levels
Description: Descriptive statistics
Time Frame: baseline and 6 months
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Aspirin
Number analyzed (Participants) | 4
pg/mL | 1.42 [0.23 to 1.98]

ADVERSE EVENTS:
Arm/Group | Aspirin
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No